CLINICAL TRIAL: NCT03003026
Title: Bike Skills Training for Children With Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Bike Skills Training for Children With Cerebral Palsy
Acronym: CPBIKERCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Melbourne (Other); Deakin University (Other); Monash Medical Centre (Other)
Responsible Party: Principal Investigator, Rachel Toovey, PhD candidate | Physiotherapist, Murdoch Childrens Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36209; S16-007 (Other Grant/Funding Number: Physiotherapy Research Foundation); HREC/116/RCHM/16 (Other: Multisite HREC ID); RES-16-0000555X (Other: Monash Health site specific ID)
Record Dates: First submitted 2016-12-04; First posted 2016-12-26 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Palsy
Keywords: motor learning; participation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel task-specific program (Experimental): Intervention arm - see detailed intervention group description below
  Interventions: Other: Novel task-specific bike skills training program
- Parent-led home-based program (Active Comparator): Comparison arm - see detailed comparison group description below
  Interventions: Other: Parent-led home-based bike skills training program

INTERVENTIONS:
Other: Novel task-specific bike skills training program — Participants randomised to the intervention group will participate in a novel task-specific bike skills training program. The intervention involves seven key components: it is group-based, intensive (2 hours per day for 3 days plus a home program for the remaining days of the one week period), task-specific, goal-directed, and therapist led, with parent involvement and conducted in an ecological setting. Each program will be run by a physiotherapist and allied health assistant during the school holidays.
  Arms: Novel task-specific program
Other: Parent-led home-based bike skills training program — The comparison group will involve a parent-led home-based bike skills training program. Parents of children randomized to the comparison group will receive written information and telephone support from a physiotherapist on training bike skills. They will be encouraged to work with their child towards their bike skills goals for at least 30-45 minutes per day over a one week period during the school holidays in home and community environments.
  Arms: Parent-led home-based program

SUMMARY:
An assessor blinded multi-centre randomized controlled trial will be conducted in which 60 participants will be randomized to either a novel task-specific approach to training bike skills or a parent-led home program comparison group. Baseline assessment will take place within 6 weeks prior to starting the intervention (T0) and outcomes will be assessed within a week following (T1); and at 12 - 14 weeks following (T2) the week long intervention. The primary outcome is attainment of individualised two-wheel bike specific goals at T1. All statistical analysis will be conducted on an intention-to-treat basis. Logistic regression will be used to assess the effect of providing the novel intervention compared to the parent-led home program on bike-specific goal attainment.

ELIGIBILITY:
Inclusion Criteria:

* Live in Victoria, Australia
* Diagnosis of cerebral palsy
* Aged 6 - 15 years
* Independently ambulant without mobility aids
* Have goals specific to two-wheel bike skills
* Have medical clearance to participate
* Have access to an appropriate bike and helmet
* Have a primary care giver who understands written and spoken English available to participate for each participant.

Exclusion Criteria:

* Has a moderate to severe intellectual impairment
* Has a dual diagnosis with another developmental disability or medical condition that may impact on their ability or safety to train two-wheel bike skills. This includes; Autism Spectrum Disorder, Trisomy 21, spina bifida, uncontrolled epilepsy, significant visual or hearing impairment as determined by medical clearance from the child's general practitioner or paediatrician
* Had musculoskeletal surgery, or other major surgery including insertion of a baclofen pump that may affect their physical ability, in the 6 months prior to randomisation or during the intervention and 12 week follow up period (if after randomisation, will be excluded from per-protocol analysis)
* Has Botulinum toxin-A (BonT-A) injections to the lower limbs and/or upper limbs in the 6 months prior to randomisation, or during the intervention and 12 week follow up period (if after randomisation, will be excluded from per-protocol analysis)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Goal attainment at 1 week post the intervention period as measured by the Goal Attainment Scale (GAS) | 1 week following intervention
  The GAS is a criterion referenced tool for individualized and collaborative goal setting between the child, family and therapist. Two to three individualized goals specific to two-wheel bike riding per participant will be set at the baseline visit with six potential outcomes specified for each goal from (-3 (deterioration), -2 (equal to start), -1 (less than expected), 0 (expected), 1 (somewhat more than expected), 2 (more than expected)). For each goal, attainment is defined as a score of zero or above on the GAS. The primary outcome, goal attainment, will be defined as attainment of at least one goal to an expected (score of zero) or greater level.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Toovey, PT, MPH, Principal Investigator — Murdoch Childrens Research Institute
Locations (2):
- Australia (2):
  - Monash Health, Clayton, Victoria
  - The Royal Children's Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toovey R, Harvey AR, McGinley JL, Lee KJ, Shih STF, Spittle AJ. Bike skills training for children with cerebral palsy: protocol for a randomised controlled trial. BMJ Open. 2018 Feb 3;8(2):e019898. doi: 10.1136/bmjopen-2017-019898. PMID 29431140